CLINICAL TRIAL: NCT00253136
Title: Risperidone Depot (Microspheres) vs. Placebo in the Treatment of Subjects With Schizophrenia
Brief Title: A Study of the Effectiveness and Safety of Long-acting Injectable Risperidone Versus Placebo in the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006055
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: schizophrenia; schizoaffective disorder; psychotic disorder; risperidone; long-acting injectable; intramuscular injection; antipsychotic agents
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to compare the effectiveness and safety of a long-acting injectable formulation of risperidone (an antipsychotic medication) versus placebo for the treatment of the symptoms of schizophrenia over a 12-week period.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that causes changes in a person's perception, thoughts, and behaviour. In schizophrenics, the most common symptoms are positive symptoms (delusions and hallucinations), negative symptoms (avoiding social situations, lack of feeling or expression), and disorganized symptoms (confusion in thinking and speech). Because of the serious nature of these diseases, it is important that patients with schizophrenia take their antipsychotic medication regularly. Long-acting injectable forms of antipsychotic drugs may eliminate the need for daily oral medication and increase a patient's compliance in taking their medication as prescribed by their physician. This is a randomized, double-blind, parallel-group, placebo-controlled study comparing the effectiveness and safety of an injectable formulation of risperidone (coated microspheres) to placebo in patients with schizophrenia. The study is composed of two periods: a 1-week run-in period (patients discontinue other antipsychotic drugs and receive oral risperidone, up to 4 mg/day) and a 12 week double-blind period during which subjects are randomized to receive bi-weekly injections of placebo or risperidone long-acting injectable formulation (25, 50, or 75 mg). During the first 3 weeks of double-blind treatment, patients will receive supplemental daily oral doses of placebo or risperidone tablets. The primary measure of effectiveness is the change from baseline in the total score for the Positive and Negative Syndrome Scale for Schizophrenia (PANSS). The PANSS is a rating scale that measures the symptoms of schizophrenia. Safety evaluations include the incidence of adverse events, results of clinical laboratory tests (hematology, biochemistry, urinalysis), measurements of vital signs and body weight, physical examination and electrocardiogram (ECG) findings, clinical examination of the injection area (buttocks), and the Extrapyramidal Symptoms Rating Scale (ESRS), a scale used to measure effects of antipsychotic medications on motor functions of the patient. Additional testing conducted includes the Clinical Global Impressions (CGI), a rating system used to evaluate the overall and severity of clinical change in a patient with various diseases affecting the brain, and the SF-36 Health Survey, a questionnaire the patient fills out that is extensively used to rate a patient's quality of life. The study hypothesis is that the injectable form of risperidone will be more effective than placebo, as measured by the change from baseline in the total PANSS score, in patients with schizophrenia. 1-week run-in period: risperidone oral tablets, up to 4 mg/day. During the first 3 weeks of double-blind period: risperidone oral tablets, 2, 4, or 6 mg/day or placebo tablets. Day 1 of double-blind period and every 2 weeks thereafter: risperidone intramuscular injection (25, 50, or 75 mg) or placebo injection for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, according to the Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV) criteria
* total score at study entry on the PANSS (Positive and Negative Syndrome Scale for Schizophrenia) of >=60 and <=120
* patient is otherwise healthy on the basis of a pre-trial physical examination, medical history, electrocardiogram (ECG) findings and results of clinical hematology, biochemistry, and urinalysis tests performed within 1 week of the start of risperidone treatment
* women of child-bearing age must be using an adequate method of birth control and have a negative pregnancy test before the start of risperidone treatment.

Exclusion Criteria:

* Patients receiving an injectable form of another antipsychotic (last injection within 120 days of screening)
* patients with a DSM-IV Axis I diagnosis other than schizophrenia
* DSM-IV diagnosis of substance dependence within 3 months of start of screening (nicotine and caffeine dependence are allowed)
* history or current symptoms of tardive dyskinesia (a condition seen in patients receiving long-term medication with certain types of antipsychotics in which the patients develop movements of the tongue, lips, face, trunk and hands and feet that they cannot control)
* history of neuroleptic malignant syndrome (a rare condition in patients receiving antipsychotic medication in which a patients may develop fever, sweating, unstable blood pressure, rigid muscles, and other symptoms, including changes in their normal mental state).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 458 (Actual)
Dates: Start 1999-11; Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of double-blind treatment in the PANSS (Positive and Negative Syndrome Scale for Schizophrenia) total score

SECONDARY OUTCOMES:
PANSS subscale scores; CGI (Clinical Global Impressions) scores and change from baseline in CGI; SF-36 (Quality of Life) evaluations; safety evaluations conducted throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- [Result] Kane JM, Eerdekens M, Lindenmayer JP, Keith SJ, Lesem M, Karcher K. Long-acting injectable risperidone: efficacy and safety of the first long-acting atypical antipsychotic. Am J Psychiatry. 2003 Jun;160(6):1125-32. doi: 10.1176/appi.ajp.160.6.1125. PMID 12777271